CLINICAL TRIAL: NCT02271022
Title: Utilization of Ticagrelor in the Upstream Setting for Non-ST-Segment Elevation Myocardial Infarction (UPSTREAM): An ED-Based Clinical Registry
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-BRIL-UPSTREAM
Record Dates: First submitted 2014-10-10; First posted 2014-10-22 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Acute Coronary Syndromes
Keywords: ACS, Acute Coronary Syndromes; NSTEMI; MI, Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Patients (≥18 years of age) with a working diagnosis of NSTEMI and treatment with an OAP agent (ticagrelor, clopidogrel, or prasugrel) either in the ED, or in any case within the timeframe that emergency physicians consider to be "upstream"-within the first 72 hours of care and at least 4 hours before diagnostic angiography. In addition, only those patients who undergo a diagnostic coronary angiography within 72 hours of ED arrival will be eligible for UPSTREAM.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
The primary objective of the UPSTREAM Registry is to address the data gap regarding the course of NSTEMI (Non-ST-Elevation Myocardial Infarction)between ED (Emergency Department) arrival and diagnostic angiography in detail, by characterizing and following the ED and peri-ED use of advanced OAP (Oral Anti-Platelet) agents. In addition to exploring ED treatment patterns and success of both ischemic and bleeding risk stratification prior to definition of the coronary anatomy, data generated via the UPSTREAM registry will allow plausible attribution of ischemic and bleeding outcomes to pre-catheterization antiplatelet therapy in the management of NSTEMI. This registry further seeks to demonstrate that contemporary use of upstream ticagrelor is associated with an economically-sound utilization of hospital resources, and smooth transition of care into the outpatient, secondary prevention setting for the first 30 days after hospitalization. Finally, it will allow characterization of patient selection factors and processes for ticagrelor vs alternative OAP agents, carrying out that descriptive comparison through discharge. Patients transferred in to an UPSTREAM hospital are eligible for inclusion, but the timing for OAP agent administration and diagnostic catheterization begin with ED care at the first hospital.

DETAILED DESCRIPTION:
This is a Phase IV, post-approval, multicenter, prospective, noninterventional study of consecutive patients with a working diagnosis of NSTEMI (Non-ST-Elevation Myocardial Infarction) and treatment with an OAP (Oral Anti-Platelet) agent (ticagrelor, clopidogrel, or prasugrel) either in the ED (Emergency Department), or in any case within the timeframe that emergency physicians consider to be "upstream"- i.e., within the first 72 hours after ED arrival and at least 4 hours before diagnostic angiography. This registry is designed to address the data gap regarding the course of NSTEMI between ED arrival and diagnostic angiography in detail, by characterizing and following the ED and peri-ED use of advanced OAP agents.

Demographic, ischemic vs bleeding risk stratification [calculated retrospectively by GRACE (Global Registry of Acute Coronary Events), TIMI (Thrombolysis in Myocardial Infarction), and PURSUIT (Platelet glycoprotein IIb/IIIa in Unstable angina: Receptor Suppression Using Integrilin) scores, and CRUSADE (Can Rapid risk stratification of Unstable angina patients Suppress ADverse outcomes with Early implementation of the ACC/AHA guidelines) Bleeding Score, respectively], and OAP agent data (including, when discernible, rationale for agent selection) will be collected for all UPSTREAM patients, regardless of OAP therapy, through discharge. Risk factors, angiography results, intervention/s (if any), post-catheterization care, discharge regimens, and in-hospital outcomes will be recorded.

Patients who are treated upstream, in-hospital, and are discharged home on ticagrelor, will be further followed up, by telephone and/or chart review (if necessary elements are included in chart accessible to investigator), at 30 (+10) days post-discharge, during which evaluation data elements to be collected include patient-reported compliance with visits and medications, patient-reported healthcare resource utilization, and any pertinent events or complications.

Patients who are treated upstream, in-hospital, or discharged home on a different OAP therapy (clopidogrel or prasugrel) will not be followed beyond the data collection completed at hospital discharge. It is expected that a relatively small number of patients will change therapy from ticagrelor to another OAP agent after discharge and prior to 30 days post-discharge, though such changes will be queried in the 30-day call/chart review.

ELIGIBILITY:
Inclusion Criteria:

Patients (≥18 years of age) with a working diagnosis of NSTEMI and treatment with an OAP agent (ticagrelor, clopidogrel, or prasugrel) either in the ED, or in any case within the timeframe that emergency physicians consider to be "upstream"- i.e., within the first 72 hours of care and at least 4 hours before diagnostic angiography. In addition, only those patients who undergo a diagnostic coronary angiography within 72 hours of ED arrival will be eligible for UPSTREAM.

Exclusion Criteria:

1. Life expectancy less than 90 days in opinion of treating clinician;
2. Not undergoing diagnostic angiography within 72 hours of ED arrival;
3. Refusal of consent; or
4. Unlikely to comply with follow-up by telephone.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (≥18 years of age) with a working diagnosis of NSTEMI and treatment with an OAP agent (ticagrelor, clopidogrel, or prasugrel) either in the ED, or in any case within the timeframe that emergency physicians consider to be "upstream"-within the first 72 hours of care and at least 4 hours before diagnostic angiography. In addition, only those patients who undergo a diagnostic coronary angiography within 72 hours of ED arrival will be eligible for UPSTREAM.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-02-17 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Composite and individual components of cardiovascular death, MI, and stroke | 30 days
  In patients who are treated upstream, in-hospital, and who are on ticagrelor at the end of 30-days post-discharge, composite and individual components of cardiovascular death, MI (Myocardial Infarction), and stroke, and bleeding rates will be assessed within 30 days.
Bleeding rates within 30 days | 30 days
  In patients who are treated upstream, in-hospital, and who are on ticagrelor at the end of 30-days post-discharge, bleeding occurring in-hospital will be classified according to the TIMI, GUSTO (Global Use of Strategies to Open Occluded Arteries), PLATO (PLATelet inhibition and patient Outcomes), and BARC (Bleeding Academic Research Consortium) scales; bleeding reported by the patient at 30-day follow-up will also be assessed.

SECONDARY OUTCOMES:
Choice of alternative OAP agents in either the upstream setting or after switching from upstream ticagrelor to downstream or discharge clopidogrel or prasugrel will be explored and analyzed | 30 days
  Choice of alternative OAP agents in either the upstream setting or after switching from upstream ticagrelor to downstream or discharge clopidogrel or prasugrel will be explored and analyzed.
Time between administration of first upstream OAP agent and catheterization | 30 days
  Time between administration of first upstream OAP agent and catheterization will be analyzed as a continuous variable to assess more broadly the impact of OAP treatment prior to diagnostic angiography in NSTEMI.
Healthcare Resource Utilization | 30 days
  In patients who are treated upstream, in-hospital, and who are on ticagrelor at the end of 30-days post-discharge, healthcare resource utilization data will be captured throughout the 30 day continuum.

CONTACTS AND LOCATIONS:
Overall Officials: Charles V. Pollack, MA, MD, FACEP, FAAEM, FAHA, Principal Investigator — Hospital Quality Foundation
Locations (48):
- United States (48):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Sacramento, California
  - Research Site, Bridgeport, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Peoria, Illinois
  - Research Site, Richmond, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Bloomfield, Michigan
  - Research Site, Grand Blanc, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, Camden, New Jersey
  - Research Site, Flemington, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Piscataway, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Roseburg, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, York and Ephrata, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Galveston, Texas
  - Research Site, McKinney, Texas
  - Research Site, New Braunfels, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Manitowoc, Wisconsin
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- See also: study report synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=NIS-BRIL-UPSTREAM&attachmentIdentifier=ac170880-09e2-4ccf-8819-0793f53dca5d&fileName=STUDY_REPORT_SYNOPSIS_Redacted.pdf&versionIdentifier=